CLINICAL TRIAL: NCT03488511
Title: The Impact of Preoperative FoodforCare at Home on Nutritional and Functional Outcomes
Brief Title: The Impact of Preoperative FoodforCare at Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-3043
Record Dates: First submitted 2018-03-21; First posted 2018-04-05 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-04

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive meals from FoodforCare at Home. The FoodforCare at Home concept consists of six small protein and energy enriched meals and snacks that will be delivered twice a week. After an individual intake, the composition of the dishes will be tailored to the needs of the patient in terms of composition, diet, taste, flavor and portion size. Besides the meals, patients in the intervention group will also receive an information leaflet about the importance of protein during treatment and how to reach their protein requirements.
  Interventions: Other: FoodforCare at home
- Control group (No Intervention): The control group will continue their usual diet for 3 weeks and have no restrictions to their diet.

INTERVENTIONS:
Other: FoodforCare at home — Six small protein rich meals that will be delivered twice a week for 3 weeks.
  Arms: Intervention group

SUMMARY:
Preoperative nutritional state is closely related to perioperative morbidity and complications. This study aims to determine the effect of a protein-rich meal service in the preoperative setting compared to usual care.

DETAILED DESCRIPTION:
Each year, approximately 1.4 million patients in the Netherlands are operated. Adequate nutritional intake, mainly protein intake, before surgery is important to improve preoperative muscle strength and functional capacity. However, up to 40% of patients admitted to the hospital suffer from malnutrition and this further deepened during hospitalization, which is an independent risk factor for peri-operative morbidity and severe complications, ranging from increased muscle loss, to higher infection rates, delayed wound healing and subsequently a prolonged hospital stay. An adequate food service is one strategy to improve protein intake and thereby the nutritional status. Extension of the study period to the out-of-hospital setting is recommended to explore the effects of long-term exposure to this concept on nutritional, functional and clinical outcomes. Therefore, the investigators aim to evaluate whether home delivered protein-rich meals, as part of FoodforCare meal service, in the preoperative setting improves protein intake in patients undergoing surgery, compared to usual care. The second aim is to investigate the effects on functional and clinical outcomes.

ELIGIBILITY:
Inclusion criteria:

* 18 years or older
* surgical patients
* living within a 40 km radius around Nijmegen/Veghel
* inclusion at least 4 weeks before surgery
* surgery: Urology, Orthopedics, Gynaecology, General Surgery
* oral intake

Exclusion criteria:

* renal insufficiency (MDRD-GFR (glomerular filtration rate) < 60ml/min and/or proteinuria)*
* food allergy
* planned vacation during intervention period

  * proteinuria is defined in case of a protein creatinine ratio > 0.5g/10mmol or an albuminuria > 300mg/day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Protein intake relative to requirements | 3 weeks
  3-day food diary filled in at baseline and after 3 weeks.

SECONDARY OUTCOMES:
Nutritional status | 3 weeks
  Patient Generated Subjective Global Assessment (PG-SGA) performed at baseline and after 3 weeks.
Quality of life and overall health status | 3 weeks
  ShortForm-36 questionnaire filled in at baseline and after 3 weeks. This questionnaire consists of 36 questions about physical and psychological aspects. Each item is scored on a 0 to 100 range. The higher the score, the higher the quality of life of the patient.
Patient satisfaction | 3 weeks
  Questionnaire filled in after 3 weeks of receiving meals. This is a self-developed questionnaire which does not have a total score. Each question will be analyzed separately. Questions consist of grading from 0-10 (the higher, the better the outcome) or with a 5-point Likert scale (completely disagree-completely agree).
Length of stay | 2 months
  These are determined retrospectively in the electronic patient file EPIC 2 months after baseline
Readmissions | 2 months
  These are determined retrospectively in the electronic patient file EPIC 2 months after baseline
Postoperative complications | 2 months
  This is reported using a standardized classification system 2 months after baseline
Energy intake relative to requirements | 3 weeks
  3-day food diary filled in at baseline and after 3 weeks.
Functional status | 3 weeks
  Short Physical Performance Battery (SPPB) performed at baseline and after 3 weeks.
Muscle strength | 3 weeks
  Hand grip strength (kg) performed at baseline and at 3 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Manon van den Berg, PhD, Study Chair — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Maasziekenhuis Pantein, Beugen, North Brabant

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-02): https://cdn.clinicaltrials.gov/large-docs/11/NCT03488511/Prot_SAP_000.pdf